CLINICAL TRIAL: NCT06925204
Title: Natural Course and Therapeutic Effect of Chronic Pancreatitis: a Prospect Cohort Study
Brief Title: Natural Course and Therapeutic Effect of Chronic Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: CCPC
Record Dates: First submitted 2025-03-20; First posted 2025-04-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patient's stool, blood, urine, pancreatic tissue and pancreatic stones generated during the diagnosis and treatment will be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic pancreatitis: This group included all enrolled patients with CP.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Based on the patient's specific clinical condition, the appropriate examination and treatment in accordance with the conventional diagnosis and treatment standards of CP will be performed, including but not limited to: CT, MRI, endoscopic ultrasound (EUS) with or without biopsy, endocrine hormone testing (such as oral glucose tolerance test or mixed meal tolerance testing), pancreatic exocrine function tests (such as fecal elastase-1 test), extracorporeal shock wave lithotripsy (ESWL), endoscopic retrograde cholangiopancreatography (ERCP), and pancreatic enzyme replacement therapy. Patients were followed up regularly.

SUMMARY:
The goal of this observational study is to establish a prospective cohort of chronic pancreatitis (CP) patients to provide evidence-based guidance for clinical practice and comprehensively optimize diagnostic and treatment strategies. The study aims to collect detailed demographic information, clinical data, medical imaging, biological samples, and follow-up information from CP patients.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is clinically characterized by abdominal pain and pancreatic dysfunction, including diabetes and steatorrhea, which significantly impact patients' quality of life and life expectancy. Globally, the annual incidence of CP is 9.62 per 100,000 individuals, with a mortality rate of 0.09 per 100,000 and a prevalence ranging from 13.5 to 560 per 100,000. In China, the prevalence of CP has also been increasing annually, currently reaching 13.52 per 100,000 individuals. In most countries worldwide, the incidence and prevalence of CP are generally on the rise, leading to an increasing healthcare burden. Due to the endocrine and exocrine functions of the pancreas, CP presents with highly variable clinical symptoms, diverse complications, and a risk of malignant transformation. Therefore, establishing a standardized, large-scale, long-term follow-up prospective cohort for CP is crucial for a more comprehensive understanding of its clinical characteristics and for providing high-quality evidence-based medical guidance for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic pancreatitis.

Exclusion Criteria:

* Patients who refuse to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic pancreatitis patients in China.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2035-12-01 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | Annually for 10 years post-enrollment (Year 1 through Year 10)
  The incidence of complications after the diagnosis of chronic pancreatitis, including diabetes mellitus, pancreatic exocrine insufficiency, pancreatic pseudocyst, biliary stricture, pancreatic portal hypertension, and pancreatic fistula.

SECONDARY OUTCOMES:
Incidence of pancreatic cancer | 5 and 10 years after enrollment
  The incidence of pancreatic cancer after the diagnosis of chronic pancreatitis
Efficacy of endoscopic treatment | 1 year after treatment
  Proportion of patients with chronic pancreatitis who had pain relief after conservative, endoscopic (ESWL and ERCP), or surgical treatment
Scores of quality of life | Annually for 10 years post-enrollment (Year 1 through Year 10)
  Quality of life scores for patients with chronic pancreatitis are obtained using SF-36 (36-Item Short Form Health Survey) which contains 8 dimensions scored from 0 to 100 (standardized converted scores). The higher score means better function.
HbA1c level | Baseline and Year 1 to Year 10 post-enrollment (annually)
  Glycated hemoglobin (HbA1c) level measured in venous blood (unit: %).
Blood glucose profile characteristics | Baseline and Year 1 to Year 10 post-enrollment (annually)
  Blood glucose profile from mixed-meal glucose tolerance test (MMTT) and continuous glucose monitoring system (CGMS) (unit: mmol/L or mg/dL).
Pancreatic and gut hormone levels | Baseline and Year 1 to Year 10 post-enrollment (annually)
  Levels of specific pancreatic hormones (C-peptide, insulin, glucagon, etc.) and gut hormones (ghrelin, gastric inhibitory peptide, glucagon like peptide-1, etc.) measured in venous blood (unit: specify for each hormone).

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kichler A, Jang S. Chronic Pancreatitis: Epidemiology, Diagnosis, and Management Updates. Drugs. 2020 Aug;80(12):1155-1168. doi: 10.1007/s40265-020-01360-6. PMID 32647920
- [Result] Oh TK, Song IA. Five-year mortality trends associated with chronic pancreatitis in South Korea: A population based cohort study. Pancreatology. 2020 Jul;20(5):828-833. doi: 10.1016/j.pan.2020.04.024. Epub 2020 Jun 18. PMID 32646739
- [Result] Sellers ZM, MacIsaac D, Yu H, Dehghan M, Zhang KY, Bensen R, Wong JJ, Kin C, Park KT. Nationwide Trends in Acute and Chronic Pancreatitis Among Privately Insured Children and Non-Elderly Adults in the United States, 2007-2014. Gastroenterology. 2018 Aug;155(2):469-478.e1. doi: 10.1053/j.gastro.2018.04.013. Epub 2018 Apr 13. PMID 29660323
- [Result] Wang LW, Li ZS, Li SD, Jin ZD, Zou DW, Chen F. Prevalence and clinical features of chronic pancreatitis in China: a retrospective multicenter analysis over 10 years. Pancreas. 2009 Apr;38(3):248-54. doi: 10.1097/MPA.0b013e31818f6ac1. PMID 19034057